CLINICAL TRIAL: NCT05488977
Title: The Effects of Endurance Training in Women With Lipedema
Brief Title: The Effects of Endurance Training on Lipedema
Acronym: LipidEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 461077
Record Dates: First submitted 2022-07-08; First posted 2022-08-05 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Lipedema
MeSH Terms: conditions — Lipedema | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training (Experimental): 8 weeks of supervised high-intensity interval training (HIIT) that is 4×4 min intervals at 85-95% of maximal heart rate (HRmax) with 3-minute active breaks (~60 % HRmax) in between intervals, twice a week) on treadmills. In addition, the participants will perform exercise once a week on their own following the correct exercise intensity.
  Interventions: Behavioral: Exercise training
- Control (No Intervention): No intervention. Carry on their normal life.

INTERVENTIONS:
Behavioral: Exercise training — 8 weeks of supervised high-intensity interval training (HIIT).
  Arms: Exercise training

SUMMARY:
Lipedema is a fat disorder causing accumulation of subcutaneous adipose tissue particularly in arms and legs, and predominantly affects women. Lipedema likely contributes to an array of other pathologies, including obesity, inflammatory bowel disease, and neurological disorders. Lipedema tissue is often very painful and can severely impair mobility. The condition can also increase the incidence of depression, anxiety, or eating disorders.

There seems to be a general impression that lipedema tissue is difficult to reduce by diet, exercise, or bariatric surgery. However, only a few studies have actually explored the effects of exercise training on lipedema. Despite the lack of knowledge, the existing guidelines for lipidemia treatment promote a healthy lifestyle with individually adjusted weight control measures, including physical activity. In general, exercise is known to have an important effect on adipose tissue. Excess adipose tissue causes macrophage infiltration into the adipose tissue leading to continuous low systemic inflammation. This would suggest that there is a systemic inflammatory response in lipedema patients. Increasing IL-6 levels with exercise can decrease the level of proinflammatory TNFalpha synthesized from adipocytes and therefore lead to an anti-inflammatory effect by increasing IL-10 and IL-1ra levels. IL-6 also stimulates fat oxidation by increasing lipolysis. For these reasons, adding an appropriate exercise program to standard treatment might provide additional benefits for lipedema patients. The investigators aim to determine the therapeutic potential of high-intensity interval training (HIIT) on pain, quality of life, body composition, cardiorespiratory fitness and circulating biomarkers in women with lipedema.

DETAILED DESCRIPTION:
Methods

Subjects 30 women diagnosed with lipedema age 18-65 will be randomized to (1:1) to 8 weeks of exercise training og a control group. Exclusion criteria includes ongoing eating disorders and/or orthopedic limitations for exercise training. A compliance with the training program of 80% will also be set as a criterion for completing the study. Participants will be recruited via social media, via physiotherapists, via posters at GPs and via a user representative from the Norwegian Lymphedema and Lipedema Association (NLLF). The master's students will obtain informed consent cf. GCP and the Health Research Act. The potential participants will have at least one week to consider their participation. If a research participant should be injured on the basis of something the investigators ask them to do, NTNU will have the insurance responsibility. The investigators will collect data on the type and stage of lipedema, when the participant was diagnosed. The investigators will also collect data on which clinical aids they are using and how often, e.g., compressions aids.

Intervention - Training protocol The women will be randomized (1:1) to 8 weeks of supervised high-intensity interval training (HIIT) that is 4×4 min intervals at 85-95% of maximal heart rate (HRmax) with 3-minute active breaks (~60 % HRmax) in between intervals, twice a week) on treadmills at the NextMove core facility at NTNU or to a control group. All participants will be provided with a pulse watch to keep after the study is completed. In addition, the participants will perform exercise once a week on their own following the correct exercise intensity. Pool training will be recommended based on potential benefits from compression. Body composition, blood pressure, VO2max (maximal oxygen uptake), questionnaire data and blood samples will be measured/collected before and after the exercise intervention. The participants will write a diary for their physical activity using standardized templates from the NextMove core facility.

Maximal oxygen uptake (VO2max) VO2max will be measured during uphill treadmill walking or running (Woodway PPS 55 Med, Munich, Germany), using ergospirometry (Jaeger, Oxycon pro, Hoechberg, Germany / Meta Max II, Cortex, Leipzig, Germany) as described earlier.11 A warm-up period for 10 min (~60% of HRmax) will precede the test. A levelling off of oxygen uptake (VO2) despite increased work load and respiratory exchange ratio ≥1.05 will be used as criteria for VO2max. HR will be measured continuously during the test (Polar, Polar Electro, Kempele, Finland), to define HRmax.

Anthropometric measurements Body weight, body mass index and waist-to-hip ratio will be measured. Body composition will be measured using InBody. For measurement of body composition, the investigators will use an instrument called Inbody 720 (Body Analysis AS). Inbody 720 provides weight, muscle mass, fat percentage, metabolism and mineral status non-invasively by sending weak electrical signals through the body. The whole test lasts just a few minutes. Before the analysis the participants should be fasten at least two hours and should avoid strenuous exercise. The standard procedures at NextMove will be used to measure the weight and height of participants. The height will be measured without shoes or head wear, this must be done with equal weight on both legs. The distance between the legs shall be a foot. The heels should be in the ground at full stretch their legs. The height is measured with one decimal. The weight is measured without heavy clothes and shoes, while the participants are standing still. It will be drawn 0.5 kg for the remaining clothes. The weight is measured with one decimal. The participants must stand upright for measuring of waist and hip circumference and a regular exhaust measuring the circumference one cm over the navel. The waist circumference is measured with no decimals.

Blood pressure Blood pressure will be measured while the patient is sitting down and have been resting for at least five minutes in a quiet room. It will be measured by a trained person, with a handheld sphygmomanometer (Tycos, 5098-02CB, USA). Blood pressure will be measured at the same time of the day for each individual at pre- and post test. The first reading will be discarded and the mean of the next three consecutive readings with a coefficient of variation below 15% will be used in the study, with additional readings if required. The sleeve should be placed at heart level and customized with the size of the participants arm.

Pain and fatigue registration Visual analog scale (VAS), measured by means of a 0-100 mm, for pain will be used to collect data on pain. VAS has been used in the social and behavioral sciences to measure a variety of subjective phenomena. A VAS is a straight line, whose end anchors indicate the extreme boundaries of the sensation, feeling, or responses to be measured. For example a VAS to measure pain can be labeled "no pain" on one end and "pain as bad as it could possibly be" on the other end. Subjects respond to the VAS by placing a mark through the line at a position which best represents their current perception of a given phenomenon between the labeled extremes. Although a VAS may be horizontal or vertical and of any length deemed appropriate, its most common form is a 100 mm horizontal line. The VAS is scored by measuring the distance, usually in millimeters, from one end of the scale to the subject's mark on the line. In the present study, a score from 1-100 was used for measuring self reported total pain and fatigue. LYMQOL (Lymphoedema Quality of Life) BEN and Brief Pain Inventory will be applied.

Quality of life questionnaires Short Form Health Survey-36 (SF-36) will be used to track potential changes in quality of life. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The eight sections are; vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health.

Standard blood analyses Blood collection and blood analyses will be performed using standard local procedures for the general biomarkers in clinical use and will be performed in all participants at the pre- and post-test. Three 3ml EDTA-tubes and one 3ml Li-heparin-tube will be collected and sent to clinical-chemical analyses at St.Olav's hospital. Parameters to be analyzed includes e.g. glucose, HbA1C, triglycerides, HDL-cholesterol, total cholesterol, serum ferritin and hs-CRP. An additional two tubes of blood (serum and EDTA) will be collected for later explorative biomarker assays. These blood samples will be centrifuged and aliquoted before freezing and storing in the LipidEx-biobank. A test from the standard laboratory that is without normal range may indicate a need for following up by a doctor, will be reported back to the participant as soon as possible, thus they will be asked to contact their general practitioner. The participants must fast at least three-hours before blood sampling. The time of last meal time for participants will be recorded on the patient form.

ELISA for lipedema biomarkers The ELISA technique can detect an amount of a given protein, antibody, or antigen in a sample. Explorative biomarkers outside clinical use will be assayd by ELISA methods established at the local laboratories at the Department of Circulation and Medical imaging. Potential biomarkers include TNFalpha, interleukines as well as PF4/CXCL4.

NMR Lipidomics/metabolomics/inflammatomics To explore the beneficial effects of HIIT on blood profile in these individuals, NMR (nuclear magnetic resonance) technology will be applied to determine if changes occur on the 1) lipoprotein subfractions that cannot be detected by measuring standard lipids, 2) changes occur in the metabolome and 3) changes occur in the inflammatory status. Lipidomics is a recently developed research area that apply different techniques to perform large-scale analyses of circulating lipids. NMR lipidomics utilizes differences in lipoprotein composition, size and density to extract information on lipoprotein subclasses. Several studies have demonstrated an association between lipoprotein subfractions and future cardiovascular health. This suggest that more refined analyses of lipoprotein subfractions may lead to further improvements in monitoring cardiovascular health. Lipidomics technology has developed rapidly over the past decade, to the point where clinical application now is possible.

Statistical power This is a pilot study, as there is very limited knowledge on exercise as treatment for lipedema. That is, no variables are available for power calculations. The investigators have chosen to set the number to 15 in each group to be able to account for up to 20% drop-outs. With the limited time available during a Master's project, this is a realistic target.

Data protection Patient information will be stored and handled in conformity with Norwegian laws and regulations.

ELIGIBILITY:
Inclusion Criteria:

- can meet for supervised exercise training in Trondheim.

Exclusion Criteria:

* eating disorders and/or orthopedic limitations for exercise training

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | Change from baseline to 8 weeks
  Visual analog scale (VAS), measured by means of a 0-100 mm, for pain will be used to collect data on pain. VAS has been used in the social and behavioral sciences to measure a variety of subjective phenomena. A VAS is a straight line, whose end anchors indicate the extreme boundaries of the sensation, feeling, or responses to be measured. For example, a VAS to measure pain can be labeled "no pain" on one end and "pain as bad as it could possibly be" on the other end. Subjects respond to the VAS by placing a mark through the line at a position which best represents their current perception of a given phenomenon between the labeled extremes. Although a VAS may be horizontal or vertical and of any length deemed appropriate, its most common form is a 100 mm horizontal line. The VAS is scored by measuring the distance, usually in millimeters, from one end of the scale to the subject's mark on the line.

SECONDARY OUTCOMES:
LYMQOL (Lymphoedema Quality of Life) legs | Change from baseline to 8 weeks
  Self-reported questionnaire reporting quality of life adapted to lipedema patients.
  This questionnaire has been designed and validated for patients with chronic oedema/ lymphoedema of one or both legs to measure quality of life. The patients will tick the box that best describes how they feel about each of the questions.The questionaire includes 22 main questions. The patient may tick one of the following; "Not at all", "A little", "Quite a bit" or "A lot". The last question includes a scale. The title of the scale is "Overall, how would you rate your quality of life at present?". The minimum value is 0 and mean Poor, whereas the maximum value is 10 and means Excellent.
Brief Pain Inventory | Change from baseline to 8 weeks
  Self-reported questionnaire reporting pain. The Brief Pain Inventory is a validated, widely used, self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions. The title of the scale is pain. The BPI scale defines pain as follows:
  Worst Pain Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain.
Short Form Health Survey-36 (SF-36) | Change from baseline to 8 weeks
  Self-reported questionnaire reporting quality of life. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Glucose | Change from baseline to 8 weeks
  Serum levels of glucose
HbA1C | Change from baseline to 8 weeks
  Serum levels of HbA1C
Triglycerides | Change from baseline to 8 weeks
  Serum levels of triglycerides
HDL-cholesterol | Change from baseline to 8 weeks
  Serum levels of HDL-cholesterol
Total cholesterol | Change from baseline to 8 weeks
  Serum levels of total cholesterol
Ferritin | Change from baseline to 8 weeks
  Serum levels of ferritin
hs-CRP | Change from baseline to 8 weeks
  Serum levels of hs-CRP
Interleukin | Change from baseline to 8 weeks
  Serum levels of interleukin
PF4/CXCL4 | Change from baseline to 8 weeks
  Serum levels of PF4/CXCL4
TNFalpha | Change from baseline to 8 weeks
  Serum levels of TNFalpha
Protein levels in blood | Change from baseline to 8 weeks
  Aprox. 200 proteins will be quantified (mmol/l) in blood by nuclear magnetic resonance.
Systolic blood pressure | Change from baseline to 8 weeks
  Systolic blood pressure
Diastolic blood pressure | Change from baseline to 8 weeks
  Diastolic blood pressure
Body weight | Change from baseline to 8 weeks
  Body weight based on InBody 720
Muscle mass | Change from baseline to 8 weeks
  Total muscle mass and in different parts of the body based on InBody 720
Fat percentage | Change from baseline to 8 weeks
  Total fat percentage and in different parts of the body based on InBody 720
Resting metabolism | Change from baseline to 8 weeks
  Whole body resting metabolism based on InBody 720
Maximal oxygen uptake | Change from baseline to 8 weeks
  VO2max will be measured during uphill treadmill walking or running (Woodway PPS 55 Med, Munich, Germany), using ergospirometry (Jaeger, Oxycon pro, Hoechberg, Germany / Meta Max II, Cortex, Leipzig, Germany)

CONTACTS AND LOCATIONS:
Overall Officials: Øivind Rognmo, PhD, Study Director — Norwegian University of Science and Technology
Locations (1):
- Institute for Circulation and Medical Imaging, NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No